CLINICAL TRIAL: NCT04886492
Title: CorEvitas SPHERES (Synergy of Prospective Health & Experimental Research for Emerging Solutions) Registry for Neuromyelitis Optica Spectrum Disorder (NMOSD)
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: NMOSD-750
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NMO: Pts presenting to enrolling sites across the northern America are invited to enroll if eligible

SUMMARY:
This is a Prospective, observational research study for patients with NMOSD under the care of a licensed neurologist. Approximately 800 patients and 35 clinical sites in North America will be recruited to participate with no defined upper limit for either target.

DETAILED DESCRIPTION:
The objective of the registry is to create a cohort of patients with NMOSD. Data collected will be used to prospectively study the natural history of NMOSD, real-word effectiveness and safety of medications used to treat NMOSD, and drug utilization treatment patterns. Additionally, the data will be used to systematically evaluate the burden for patients with NMOSD and the impact of therapies on quality of life. This will be done through real time capture and adjudication of relapses, the standardized collection of patient-reported outcomes (PRO) and clinician-reported outcomes (ClinRO), the active evaluation of prevalent and incident comorbidities and adverse events, and the recording of medication utilization patterns.

Personal information is also collected from each consenting registry patient allowing for linkages to other public or private clinical and administrative databases, as well as to databases maintained by organizations focused on the care and treatment of NMOSD for the purposes of clinical, market, or outcomes research. This provides an opportunity to evaluate other aspects of the disease and its treatment including but not limited to clinical and drug cost-effectiveness, health care resource utilization, and patient adherence.

Consent for additional ad hoc surveys will be solicited which can allow evaluation of additional aspects of the disease impact such as care giver burden or impact of disease on productivity.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of NMOSD at the time of enrollment according to the 2015 IPND consensus diagnostic criteria for NMOSD†.
2. Age 18 years or older at the time of enrollment.
3. Willing to provide Personal Information.

Exclusion Criteria:

1. Has had a clinically confirmed NMOSD neuro-episode within the 12 weeks prior to enrollment.
2. Is participating or planning to participate in a double-blind randomized trial for an NMOSD drug. Note: Concurrent participation in another observational registry or open-label Phase 3b/4 trial is allowed.

   * All serology types (APQ4 +/- and MOG +/-) are eligible to enroll in the registry given they meet the 2015 IPND diagnostic criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled in the NMOSD Registry during regularly scheduled office visits. Selected neurologist are invited to participate as investigators in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
NMO epidemiology, presentation, natural history, management, and outcomes | A minimum of 10 years from last patient enrolled
  The major clinical outcomes include an assessment of the epidemiology of NMO; to better understand the presentation, natural history, management and outcomes.

SECONDARY OUTCOMES:
Physician reported- MFIS | every 6 months for 10 years
Physician reported-PD-Q | every 6 months for 10 years
Physician reported-EQ-5D-5L | every 6 months for 10 years
Physician reported-SF-MPQ-2 | every 6 months for 10 years
Physician reported-Pain Severity NRS | every 6 months for 10 years
Physician reported-PHQ-2 | every 6 months for 10 years
Physician reported-Caregiver status | every 6 months for 10 years
Physician reported - NMOSD Disability Index | every 6 months for 10 years
Physician reported - NEI VFQ-UI | every 6 months for 10 years
Physician reported - TSQM-9 | every 6 months for 10 years
Patient reported - EDSS-NMOSD Module | every 6 months for 10 years
Patient reported - MoCA | every 6 months for 10 years
Percentage of patients with history of comorbidities | every 6 months for 10 years
Relapse History | every 6 months for 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States